CLINICAL TRIAL: NCT01167413
Title: Frequency of Axial Spondyloarthropathy Among Patients Suffering From Fibromyalgia - Application of the ASAS Classification Criteria
Brief Title: Frequency of Axial Spondyloarthropathy Among Patients Suffering From Fibromyalgia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Jacob Ablin, MD, Director, Fibromyalgia Clinic, Institute of Rheumatology, Tel Aviv Sourasky Medical Center
Other Study IDs: TASMC-10-JA-0423-CTIL
Record Dates: First submitted 2010-01-24; First posted 2010-07-22 (Estimated); Last update posted 2010-08-06 (Estimated); Status verified 2010-01

CONDITIONS: Fibromyalgia; Ankylosing Spondylitis
MeSH Terms: conditions — Fibromyalgia; Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- FIbromyalgia Patients: Patients diagnosed as suffering from Fibromyalgia according to the ACR criteria
  Interventions: Device: Evaluation by manual Dolorimeter; Other: SIJ imaging

INTERVENTIONS:
Device: Evaluation by manual Dolorimeter — Patients will be examined by a manual Dolorimeter
Other: SIJ imaging — Patients will undergo imaging of the Sacroiliac joint by plain x-ray or MRI and sacroileitis will be documented

SUMMARY:
Fibromyalgia Syndrome (FMS) is a non - inflammatory condition characterized by the presence of chronic, widespread musculoskeletal pain and tenderness; FMS is considered to be the result of increased processing of pain by the central nervous system.

Axial spondyloarthropathy is the hallmark of Ankylosing Spondylitis (AS), an inflammatory joint disease involving the axial spine, the sacroiliac joints as well as peripheral joints.

Although FMS and AS differ vastly in their pathogenesis, a considerable clinical overlap may exist between these conditions. Both disorders typically cause chronic nocturnal back pain and disturbed sleep may accompany either condition. In addition,the investigators have previously described an increased prevalence of (secondary) FMS among female AS patients.

This overlap may have important clinical implications since the presence of comorbid FMS may lead to increased severity results on commonly used instruments in the evaluation of disease activity in AS, such as the BASDAI and BASFI .

Recently, the Assessment of Spondyloarthritis international Society (ASAS) has published updated classification criteria for axial spondyloarthropathy. These criteria, which are summarized in table 1, are based on the evaluation of patients suffering from chronic back pain with an age of onset of less than 45.

Objective:

The objective of the current study is to evaluate the prevalence of axial spondyloarthropathies among FMS patients, utilizing the new ASAS criteria.

ELIGIBILITY:
Inclusion Criteria:

Patients fulfilling American College of Rheumatology criteria for classification of Fibromyalgia:

* Widespread pain lasting over three months
* Tenderness in at least 11 of 18 points

Exclusion Criteria:

* Patients with known inflammatory joint disease prior to the study
* Patient not able to give informed consent
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited consecutively from the Fibromyalgia clinic as well as the general rheumatological clinic of the Tel Aviv Sourasky medical center.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-01 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Ankylosing Spondylitis as diagnosed according to ASAS criteria | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Jacob N Ablin, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center

REFERENCES:
- [Background] Aloush V, Ablin JN, Reitblat T, Caspi D, Elkayam O. Fibromyalgia in women with ankylosing spondylitis. Rheumatol Int. 2007 Jul;27(9):865-8. doi: 10.1007/s00296-007-0344-3. Epub 2007 May 3. PMID 17476510
- [Background] Sieper J, Rudwaleit M, Baraliakos X, Brandt J, Braun J, Burgos-Vargas R, Dougados M, Hermann KG, Landewe R, Maksymowych W, van der Heijde D. The Assessment of SpondyloArthritis international Society (ASAS) handbook: a guide to assess spondyloarthritis. Ann Rheum Dis. 2009 Jun;68 Suppl 2:ii1-44. doi: 10.1136/ard.2008.104018. PMID 19433414
- [Background] Wolfe F, Smythe HA, Yunus MB, Bennett RM, Bombardier C, Goldenberg DL, Tugwell P, Campbell SM, Abeles M, Clark P, et al. The American College of Rheumatology 1990 Criteria for the Classification of Fibromyalgia. Report of the Multicenter Criteria Committee. Arthritis Rheum. 1990 Feb;33(2):160-72. doi: 10.1002/art.1780330203. PMID 2306288